CLINICAL TRIAL: NCT03866512
Title: The Impact of Acipimox and Salbutamol Supplementation on the Development of Insulin Resistance and Anabolic Resistance During Forearm Immobilization in Healthy, Young Volunteers
Brief Title: Forearm Immobilization, Metabolic Health, and Muscle Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 250839; 209198/Z/17/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2019-02-28; First posted 2019-03-07 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acipimox ingestion during immobilization (Experimental): Oral ingestion of Acipimox during 2 days of forearm immobilization
  Interventions: Behavioral: Forearm immobilization
- B-agonist during immobilization (Experimental): Oral ingestion of salbutamol during 2 days of forearm immobilization
  Interventions: Behavioral: Forearm immobilization
- Placebo ingestion during immobilization (Placebo Comparator): Oral ingestion of a placebo 2 days of forearm immobilization
  Interventions: Behavioral: Forearm immobilization

INTERVENTIONS:
Behavioral: Forearm immobilization — Two days of forearm immobilization

SUMMARY:
The present study will investigate the impact of altered substrate availability on muscle atrophy, insulin sensitivity and muscle protein synthesis following short-term forearm immobilization

DETAILED DESCRIPTION:
Thirty-six healthy young volunteers will undergo 2 days of forearm immobilization combined with ingestion of one of two drug or placebo. Before and after immobilization, they will receive a stable isotope tracer infusion (5.5 h) combined with repeated blood and muscle sampling under insulin clamp conditions, in order to measure insulin sensitivity and muscle protein synthesis in the fasted and fed state.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-40 years of age
* Body mass index between 18 and 27

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 diabetes)
* Any diagnosed cardiovascular disease
* Hypertension (≥140 mmHg systolic and/or ≥90 mmHg diastolic)
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* Regular use of nutritional supplements
* Metallic implants
* A personal or family history of thrombosis, epilepsy, seizures or schizophrenia
* Any previous motor disorders
* Any known disorders in lipid metabolism
* Any known disorders in muscle metabolism
* Known allergy for Acipimox, beta agonist, or other substances in the tablets
* Known sensitivity for sympathomimetic drugs
* Known hypokalaemia
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Known severe kidney problems
* Pregnancy
* Unable to give consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlou Dirks, PhD, Principal Investigator — University of Exeter
Locations (1):
- Royal Exeter & Devon NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 57 participants were screened for their eligibility to taking part.
  n=6 were excluded, for the following reasons: n=5 BMI exceeding upper cut-off n=1 metabolic disease
  Of the remaining n=51, n=14 chose to not continue with the study.
  Of the remaining n=37, n=30 completed the study (n=3 data collection unsuccessful because of intravenous cannulation issues, n=4 dropped out)
Period: Overall Study
Arm/Group | Acipimox Ingestion During Immobilization | B-agonist During Immobilization | Placebo Ingestion During Immobilization
Started | 11 | 14 | 12
Completed | 10 | 11 | 9
Not Completed | 1 | 3 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Cannulation issues | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All completed participants were included in the analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Acipimox Ingestion During Immobilization | B-agonist During Immobilization | Placebo Ingestion During Immobilization | Total
Number analyzed (Participants) | 10 | 11 | 9 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 9 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (3) | 23 (4) | 23 (7) | 22 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 14
  Male | 5 | 6 | 5 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 11 | 9 | 30
Body mass index [Mean (Standard Deviation); unit: kg^m2] | 22.9 (2.7) | 24.1 (3.5) | 23.9 (2.1) | 23.7 (2.8)
Fat mass percentage [Mean (Standard Deviation); unit: percentage of body fat] | 20.9 (9.4) | 24.4 (12.1) | 25.1 (9.2) | 23.5 (10.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 117 (11) | 111 (9) | 114 (44) | 114 (10)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69 (6) | 70 (5) | 65 (6) | 68 (4)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Forearm Glucose Uptake
Description: Insulin sensitivity, measured as forearm glucose uptake, during a 30-min baseline period and hyperinsulinaemic-euglycaemic conditions
Time Frame: During the steady-state phase of the insulin clamp (i.e. last 30 min)
Population: All participants with completed data collection were included in the analysis
Measure: Mean (Standard Error); unit: Percent change in clamp FGU with immob
Arm/Group | Acipimox Ingestion During Immobilization | B-agonist During Immobilization | Placebo Ingestion During Immobilization
Number analyzed (Participants) | 10 | 11 | 9
Percent change in clamp FGU with immob | -73 (15) | 127 (134) | -95 (113)

2. Secondary Outcome: Percent Change in Muscle Protein Synthesis
Description: Percent change in muscle protein synthesis, measured as using the arteriovenous-venous method, via stable isotope tracer infusion
Time Frame: In the fasted state (30 min before starting insulin clamp), and during the steady-state phase of the insulin clamp (i.e. last 30 min)
Population: All participants who completed data collection were included in the analysis
Measure: Mean (Standard Error); unit: Percent change in clamp phenylalanine Rd
Arm/Group | Acipimox Ingestion During Immobilization | B-agonist During Immobilization | Placebo Ingestion During Immobilization
Number analyzed (Participants) | 8 | 11 | 9
Percent change in clamp phenylalanine Rd | -93 (40) | -124 (29) | -251 (145)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire study, up to 48h following the final study visit
Description: All participants were instructed to notify the PI of any adverse events that occurred during their enrollment in the study, and up to 48h following completion of the final study visit.
Arm/Group | Acipimox Ingestion During Immobilization | B-agonist During Immobilization | Placebo Ingestion During Immobilization
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 4/11 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acipimox Ingestion During Immobilization (N=10) | B-agonist During Immobilization (N=11) | Placebo Ingestion During Immobilization (N=9)
Nausea and vomiting (Product Issues) | 1 (1) | 4 (4) | 1 (1) — Nausea and vomiting at the end of the hyperinsulinaemic-euglycaemic clamp with amino acid co-infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03866512/Prot_SAP_000.pdf